CLINICAL TRIAL: NCT06785844
Title: Intra-rectal Botulinum Toxin Injection for Intractable Non-retentive Fecal Incontinence in Children - an Open Label Pilot Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Yogev Dotan, Dr Dotan Yogev, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intra-rectal Botulinum toxin
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-10

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Botulinum toxin (Experimental)
  Interventions: Drug: Botulinum Toxin A (Botox )

INTERVENTIONS:
Drug: Botulinum Toxin A (Botox ) — Botulinum Toxin injection

SUMMARY:
Background: Fecal Incontinence (FI) is a frustrating and prevalent GI condition with profound social implications and a marked effect on quality of life. Treatment options are limited for children whose FI is not secondary to constipation (overflow incontinence), and they are defined as having non-retentive fecal incontinence (NRFI). Rectal botulinum injections (RBI) have recently shown promise for the treatment of FI in adults, following a large, randomized placebo-controlled trial, but no data exists regarding efficacy in children.

Objectives: To evaluate the efficacy and safety of RBI in children with non-retentive fecal incontinence.

Methods: A prospective open-label pilot study. Children with intractable NRFI will be screened using anorectal manometry and a colonic transit study. Eligible patients will receive one course of RBI and data regarding FI frequency will be prospectively collected during a 15-week period.

Significance: New treatment options for children with intractable fecal incontinence are highly in need. The current study aims to introduce a new treatment modality into pediatric research and patient care.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-18 years old with fecal incontinence for a period greater than 6 months.
* FI frequency of ≥ 3 episodes/week.
* After appropriate medical evaluation, FI cannot be explained by another medical condition.
* Normal colonic transit study, defined as passage of 80% of markers on day
* Normal RAIR on anorectal manometry

Exclusion Criteria:

* Patients currently fulfilling rome IV criteria for functional constipation.
* Patients with evidence of fecal retention.
* Patients who had had good response to treatment for overflow incontinence.
* Absent RAIR on anorectal manometry.
* Any radiologic evidence of dochylosigmoid or distended colon.
* Any known organic condition that may affect bowel transit.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
median number of FI episodes/week at 1-month post-intervention compared to baseline | 3-months post-intervention
  median number of FI episodes/week at 1-month post-intervention compared to baseline. The median FI episodes/week will be calculated based on the 21-day diary. FI episode minimal definition: any episode of soiling requiring change of underwear/clothes/washing-up.

SECONDARY OUTCOMES:
Median number of FI episodes/week at 3-months post-intervention, compared to baseline diary. | 3-months post-intervention
Rate of patients with a 50% decrease in mean FI episodes/week compared to baseline diary. | 3-months post-intervention
Rate of patients with daily FI episodes (at least 1 episode/day) compared to baseline. | 3-months post-intervention
Mean number of complete bowel movements/week compared to baseline according to diary. | 3-months post-intervention
Parents and patient's general impression of the treatment using the following questions: "Was the treatment useful/beneficial?"; "Did the treatment improve your quality of life"? | 3-months post-intervention
Rate of RBI-associated major and minor adverse events. Patients will be questioned according to list, as well as allowed to add adverse events not listed. | 3-months post-intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rybak A, Martinelli M, Thapar N, Van Wijk MP, Vandenplas Y, Salvatore S, Staiano A, Benninga MA, Borrelli O. Colonic Function Investigations in Children: Review by the ESPGHAN Motility Working Group. J Pediatr Gastroenterol Nutr. 2022 May 1;74(5):681-692. doi: 10.1097/MPG.0000000000003429. Epub 2022 Feb 24. PMID 35262513
- [Background] Athanasakos E, Cleeve S, Thapar N, Lindley K, Perring S, Cronin H, Borrelli O, Mutalib M. Anorectal manometry in children with defecation disorders BSPGHAN Motility Working Group consensus statement. Neurogastroenterol Motil. 2020 Jun;32(6):e13797. doi: 10.1111/nmo.13797. Epub 2020 Jan 27. PMID 31989766
- [Background] Pascual-Pascual SI, Pascual-Castroviejo I. Safety of botulinum toxin type A in children younger than 2 years. Eur J Paediatr Neurol. 2009 Nov;13(6):511-5. doi: 10.1016/j.ejpn.2008.10.006. Epub 2008 Nov 25. PMID 19036619
- [Background] Halleran DR, Lu PL, Ahmad H, Paradiso MM, Lehmkuhl H, Akers A, Hallagan A, Bali N, Vaz K, Yacob D, Di Lorenzo C, Levitt MA, Wood RJ. Anal sphincter botulinum toxin injection in children with functional anorectal and colonic disorders: A large institutional study and review of the literature focusing on complications. J Pediatr Surg. 2019 Nov;54(11):2305-2310. doi: 10.1016/j.jpedsurg.2019.03.020. Epub 2019 Apr 23. PMID 31060739
- [Background] Leroi AM, Queralto M, Zerbib F, Siproudhis L, Vitton V, Amarenco G, Etienney I, Mion F, Bridoux V, Philip J, Brochard C, Damon H, Lacroix E, Gillibert A, Gourcerol G. Intrarectal injections of botulinum toxin versus placebo for the treatment of urge faecal incontinence in adults (FI-Toxin): a double-blind, multicentre, randomised, controlled phase 3 study. Lancet Gastroenterol Hepatol. 2024 Feb;9(2):147-158. doi: 10.1016/S2468-1253(23)00332-1. Epub 2023 Dec 18. PMID 38128556
- [Background] Kaul A, Garza JM, Connor FL, Cocjin JT, Flores AF, Hyman PE, Di Lorenzo C. Colonic hyperactivity results in frequent fecal soiling in a subset of children after surgery for Hirschsprung disease. J Pediatr Gastroenterol Nutr. 2011 Apr;52(4):433-6. doi: 10.1097/MPG.0b013e3181efe551. PMID 21240024
- [Background] Vriesman MH, Koppen IJN, Camilleri M, Di Lorenzo C, Benninga MA. Management of functional constipation in children and adults. Nat Rev Gastroenterol Hepatol. 2020 Jan;17(1):21-39. doi: 10.1038/s41575-019-0222-y. Epub 2019 Nov 5. PMID 31690829
- [Background] de Bruijn CMA, Safder S, Rolle U, Mosiello G, Marshall D, Christiansen AB, Benninga MA. Development of a Bowel Management Scoring Tool in Pediatric Patients with Constipation. J Pediatr. 2022 May;244:107-114.e1. doi: 10.1016/j.jpeds.2022.01.036. Epub 2022 Feb 1. PMID 35114289
- [Background] Koppen IJ, von Gontard A, Chase J, Cooper CS, Rittig CS, Bauer SB, Homsy Y, Yang SS, Benninga MA. Management of functional nonretentive fecal incontinence in children: Recommendations from the International Children's Continence Society. J Pediatr Urol. 2016 Feb;12(1):56-64. doi: 10.1016/j.jpurol.2015.09.008. Epub 2015 Oct 21. PMID 26654481
- [Background] Popescu M, Mutalib M. Bowel transit studies in children: evidence base, role and practicalities. Frontline Gastroenterol. 2021 May 10;13(2):152-159. doi: 10.1136/flgastro-2020-101719. eCollection 2022. PMID 35300467
- [Background] Lambregts AP, Nieuwhof-Leppink AJ, Klijn AJ, Schroeder RPJ. Intravesical botulinum-A toxin in children with refractory non-neurogenic overactive bladder. J Pediatr Urol. 2022 Jun;18(3):351.e1-351.e8. doi: 10.1016/j.jpurol.2022.02.007. Epub 2022 Feb 18. PMID 35283021
- [Background] Voskuijl WP, Reitsma JB, van Ginkel R, Buller HA, Taminiau JA, Benninga MA. Longitudinal follow-up of children with functional nonretentive fecal incontinence. Clin Gastroenterol Hepatol. 2006 Jan;4(1):67-72. doi: 10.1016/j.cgh.2005.10.001. PMID 16431307
- [Background] Rajindrajith S, Devanarayana NM, Benninga MA. Review article: faecal incontinence in children: epidemiology, pathophysiology, clinical evaluation and management. Aliment Pharmacol Ther. 2013 Jan;37(1):37-48. doi: 10.1111/apt.12103. Epub 2012 Oct 28. PMID 23106105